CLINICAL TRIAL: NCT02338167
Title: Prospective Academic Translational Research Network for the Optimization of the Oncological Health Care Quality in the Adjuvant and Advanced/Metastatic Setting: Health Care Research, Pharmacogenomics, Biomarkers, Health Economics
Brief Title: Praegnant Breast Cancer: Early/Advanced/Metastatic
Acronym: PRAEGNANT
Status: Recruiting | Type: Observational
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Other Study IDs: SEN-01/14
Record Dates: First submitted 2015-01-09; First posted 2015-01-14 (Estimated); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Advanced/Metastatic Breast Cancer; Breast Cancer (Early Breast Cancer)
MeSH Terms: conditions — Breast Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 60 Months
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Advanced/metastatic breast cancer: 3,500 patients with locally advanced, inoperable/metastatic breast cancer in any line of treatment (e.g. 1st, 2nd, 3rd, or ≥ 4th line).
  Interventions: Procedure: Blood sampling
- Early breast cancer: 10,000 patients with breast cancer in the neoadjuvant and adjuvant (early breast cancer) setting independent of treatment regimen.
  Interventions: Procedure: Blood sampling

INTERVENTIONS:
Procedure: Blood sampling — A blood sample will be taken during a routine blood draw

SUMMARY:
Among patients with breast cancer the subgroup of patients with metastases are considered the group of patients with the worst prognosis. Not only regard-ing therapy decisions but also with regard to quality assured healthcare and health economics this entity of patients remains a challenge.

Recently, novel advances in breast cancer therapy aim at the targeted therapy of tumor entities and identification of patients, for whom the greatest therapy benefit, and the least side effects are expected.

However molecular assessment of the patient and the tumor in the metastatic situation is not performed on a routine basis and in many cases tumor character-istics from the primary tumor are considered reliable enough to make therapy decisions for the metastatic patients. Although molecular reassessment of tu-mor characteristics from tumor material of the metastasis is recommended in national guidelines, only a minority of patients is biopsied, because of the inva-siveness of the procedure, even though biopsy related complications are reported to be rare.

With modern analytic methods from blood based biomaterial there seems to be an opportunity to correlate blood based tumor assessments with actual charac-teristics of the tumor. These include expression analysis, tumor mutation analy-sis, tumor gene copy number aberrations and others. One of the main aims of the PRAEGNANT study is therefore to establish an infrastructure for the compre-hensive analysis of tumor and metastatic molecular characteristics of the patient and the tumor.

Furthermore, health care related outcomes as well as health economics provide novel approaches for integration of patients in study conduct and health care awareness and are study aims of the PRAEGNANT study.

ELIGIBILITY:
Inclusion Criteria for the early breast cancer setting:

* Adult breast cancer patients (age ≥18 years)
* Patients with breast cancer and no evidence of distant metastases with a diagnosis not longer than 91 days before study entry
* Patients, who are able and willing to sign the informed consent form

Inclusion Criteria for the advanced/metastatic setting:

* Adult women aged ≥18 years
* Patients with the diagnosis of invasive breast cancer (in German: Mammakarzinom, as op-posed to "non-invasive"= ductales Carcinoma in situ; irrespective of status of BC, e.g. TNM, re-ceptor status etc.) and
* Patients, who are willing and able to sign the informed consent form
* Patients with metastatic or locally advanced, inoperable disease proven by clinical measures (i.e. standard imaging)

Exclusion Criteria:

* Patients who did not sign the informed consent form
* Patients, who are not eligible for observation due to non-availability and/or severe comor-bidities as evaluated by the treating physician

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 10,000 patients with breast cancer in the neoadjuvant and adjuvant (early breast cancer) setting independent of treatment regimen.
  3500 patients with locally advanced/metastatic breast cancer in any line of treatment (e.g. 1st, 2nd, 3rd, or ≥ 4th line). A patient can only participate after providing informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 13500 (Estimated)
Dates: Start 2014-06 (Actual); Primary Completion 2030-07 (Estimated); Study Completion 2030-07 (Estimated)

PRIMARY OUTCOMES:
MBC (Metastatic Breast Cancer): Discovery of biomarkers, which predict progression free survival (PFS) | PFS defined as the time to the first progression after study inclusion from the last time of progression before or at study entry
  Analyses will be done separately for each therapy line. Biomarkers include gene expression profiling of the primary tumor and the corresponding metastases, somatic mutations, germline genetic variation, epigenetic changes and miRNA variation up to a total of 500,000 biomarkers.
EBC (Early Breast Cancer): Assessment of disease free sur-vival (DFS) | up to 60 months
  DFS defined as the time to the first disease recurrence after study inclusion from time of primary diagnosis before or at study entry

SECONDARY OUTCOMES:
MBC: Assessment of overall survival (OS) | OS is defined as the time to death from the date of the last progression before or at study entry.
  OS is defined as the time to death from the date of the last progression before or at study entry.
MBC: Assessment of breast cancer specific survival (BCSS) | Time to death from the date of the last progression before or at study entry.
  BCSS is defined as the time to to death due to breast cancer from the date of the last progression before or at study entry.
MBC: Objective response | up to 60 months
  Objective response is defined as the best-documented response to the therapy started at study entry or the last therapy started before study entry.
MBC: Description of therapies used in the metastatic setting | after 60 months (after study completion)
  Therapies will be categorized and descriptive statistics will be presented.
MBC: Quality of life | Study entry and every 3 month or following a change of a therapy line(event-associated, e.g. after progression) until Month 24. Every 6 months from Month 24 until Death or withdrawal of consent
  Assessed with EORTC QlQ-C30 and Visual Analog Scala
MBC: Therapy adherence | up to 60 months
  Defined as the percentage of patients in which treat-ments which are terminated as per patients' wish or because of treatment related side effect.
MBC: Influencing Factors of Depression in patients with metastatic breast cancer | Study entry and every 3 month or following a change of a therapy line (event-associated, e.g. after progression) until Month 24. Every 6 months from Month 24 until Death or withdrawal of consent
  Depression will be assessed by patient reported questionnaires e.g. CESD-R.
MBC: Incidence of adverse events, serious adverse events will be reported. | up to 60 months
  According to NCI Common Toxicity Criteria Version 4.03.
MBC: Percentage of women, who will receive results of molecular tests undertaken in the context of the scientific objectives of this trial. | Once at end of study
  Number of patients who will receive molecular testing results compared to the total number of included patients.
MBC: Feasibility and satisfaction regarding receipt of molecular testing results (including hereditary genetic alterations) | Once at end of study
  Assessed with a physician and patient questionnaire and documentation of possible confirmatory testing for changes in therapy or eligibility for interventional clinical trial screening.
MBC: Health economics for women with metastatic and/or locally advanced, inoperable breast cancer. | Study entry and every 3 month or following a change of a therapy line (event-associated, e.g. after progression) until Month 24. Every 6 months from Month 24 until Death or withdrawal of consent
  EORTC QLQ C-30 (Version 3.0) (among others) and actu-al documented costs of diagnostic procedures, therapies, treatment of side effects and care for tumor-associated symptoms will be used to calculate health care costs, quality adjusted life years (QALY) and incremental cost effectiveness ratios (ICER) between patient groups.
MBC: Patient reported influencing factors on therapy adherence in patients metastatic and/or locally advanced, inoperable breast cancer. | Study entry and every 3 month or following a change of a therapy line(event-associated, e.g. after progression) until Month 24. Every 6 months from Month 24 until Death or withdrawal of consent
  Patient reported adherence for orally administered therapies will be assessed with suitable questionnaires.
EBC: Assessment of distant disease-free survival (DDFS) | Up to 60 months
  DDFS defined as the time to the first distant disease recurrence after study inclusion from time of primary diagnosis before or at study entry.
EBC: Quality of life | Study entry and every 3 month or following a change of a therapy line (event-associated, e.g. after progression) until Month 24. Every 6 months from Month 24 until Death or withdrawal of consent
  Assessed with EORTC QLQ C-30 (Version 3.0), EORTC QLQ-BR23 and the EQ-Visual Analog Scale (VAS)
EBC: Assessment of overall survival (OS) | OS is defined as the time to death from the date of the last progression before or at study entry.
  OS is defined as the time to death from the date of the primary diagnosis before or at study entry.
EBC: Assessment of breast cancer specific survival (BCSS) | Time to death due to breast cancer from the date of the primary diagnosis before or at study entry.
  BCSS is defined as the time to death due to breast cancer from the date of the primary diagnosis before or at study entry.
EBC: Description of therapies used in the early breast cancer setting | after 60 months (after study completion)
  Therapies will be categorized, and descriptive statistics will be presented.
EBC: Percentage of women, who will receive results of molecular tests undertaken in the context of the scientific objectives of this trial. | Once at end of study
  Number of patients who will receive molecular testing results compared to the total number of included pa-tients.
EBC: Feasibility and satisfaction regarding receipt of molecular testing results (including hereditary genetic alterations) | Once at end of study
  Assessed with a physician and patient questionnaire and documentation of possible confirmatory testing for changes in therapy or eligibility for interventional clinical trial screening.
EBC: Therapy adherence | up to 60 months
  Defined as the percentage of patients in which treat-ments which are terminated as per patients' wish or because of treatment related side effect
EBC: Health economics for women with breast cancer | up to 60 months
  EORTC QLQ C-30 (Version 3.0) (among others) and actu-al documented costs of diagnostic procedures, thera-pies, treatment of side effects and care for tumor-associated symptoms will be used to calculate health care costs, quality adjusted life years (QALY) and incre-mental cost effectiveness ratios (ICER) between patient groups.
EBC: Influencing Factors of Depression in patients with breast cancer | Study entry and every 3 month or following a change of a therapy line(event-associated, e.g. after progression) until Month 24. Every 6 months from Month 24 until Death or withdrawal of consent
  Depression will be assessed by patient reported ques-tionnaires e.g. CESD-R.
EBC: Patient reported influencing factors on therapy adherence in patients with early breast cancer. | Study entry and every 3 month or following a change of a therapy line(event-associated, e.g. after progression) until Month 24. Every 6 months from Month 24 until Death or withdrawal of consent
  Patient reported adherence for orally administered therapies will be assessed with suitable questionnaires.
EBC: Incidence of adverse events, serious ad-verse events will be reported. | up to 60 months
  NCI Common Toxicity Criteria Version 4.03.

OTHER OUTCOMES:
Correlation of the incidence of depression with germline gentic variation and therapies and gene expression from leukocytes. | Study entry and following a change of a therapy line (event-associated, e.g. after progression) up to month 60
  Depression Inventory values will be associated with blood biomarkers, single nucleotide polymorphisms and therapies.
Correlation of gene alterations (mutations and or amplifications) and gene expres-sion between primary tumor and metastatic tumor for the prediction of side effects and prognosis. | after 60 months (after study completion)
  DNA and RNA of the primary tumor will be extracted of archival formalin fixed, paraffin embedded tumor samples and analyzed mutations, mutation changes, and differentially expressed genes. Additionally, FFPE will be used for the construction of a TMA for antibody staining.
Correlation of gene alterations (mutations and or amplifications) and gene expres-sion between primary tumor, metastatic tumor and circulating tumor cells (CTCs). | Study entry and following a change of a therapy line (event-associated, e.g. after progression) up to month 60
  Circulating tumor cells (CTC) from selected patients will be analyzed for mutations and gene amplifications. Findings will be compared to mutations assessed from FFPE tumor material.
Correlation of gene alterations (mutations and or amplifications) between primary tumor, metastatic tumor and circulating tumor DNA. | after 60 months (after study completion)
  Circulating DNA (ctDNA) will be analyzed for genetic variation and compared to mutations assessed from FFPE tumor material.
Prediction of therapy response, prognosis and side effects with germline Single Nucleotid Polymorphisms | Study entry and following a change of a therapy line (event-associated, e.g. after progression) up to month 60
  Germline DNA will be used as reference for the genetic analysis of the tumor, CTCs and ctDNA. Additionally ge-nome-wide SNPs will be assessed and used for a ge-nome-wide association study.
Correlation of blood protein biomarkers with side effects, and progression. | Study entry and following a change of a therapy line (event-associated, e.g. after progression) up to month 60.
  EGFR (1068), HSP27 (pS78), IL-1a, IL-1b, IL-2, IL-6, Il-8, PAI-1, sEGFR, ERK1/2, mTOR, TNF-a, TNF-b. P1NP, CTX, Vitamin D, PTH, OPG, RANKL, Sclerostin, DKK-1.
Identification of risk factors for the development of metastatic disease in healthy women. | after 60 months (after study completion)
  Patients will be matched to a pool of controls, which are not part of the PRAEGNANT study, but which have been recruited during the same time.
Influencing Factors of Physical Activity, Mental factors and Nutrition in patients with metastatic breast cancer | Study entry and every 3 month or following a change of a therapy line(event-associated, e.g. after progression) until Month 24. Every 6 months from Month 24 until Death or withdrawal of consent
  Physical activity and nutrition will be assessed with patient reported questionnaires, e.g. IPAQ and ER2.
Time to progression from the beginning of subsequent therapy lines until the next progression. | up to 60 months
  All molecular and other measures that might predict prognosis will be associated with the-se times to progression as well.
Time to death from the beginning of subsequent therapy lines | up to 60 months
  All molecular and other measures that might predict prognosis will be associated with these times to death as well.

CONTACTS AND LOCATIONS:
Overall Officials: Diethelm Wallwiener, Prof. Dr., Principal Investigator — Universitätsfrauenklinik Tübingen; Peter Fasching, Prof. Dr., Principal Investigator — Frauenklinik des Universitätsklinikums Erlangen; Sara Brucker, Prof. Dr., Principal Investigator — Universitätsfrauenklinik Tübingen; Hans Tesch, Prof. Dr., Principal Investigator — Hämatologisch-Onkologische Gemeinschaftspraxis am Bethanien-Krankenhaus Frankfurt; Andreas Schneeweiss, Prof. Dr., Principal Investigator — Nationales Centrum für Tumorerkrankungen (NCT) Sektion Gynäkologische Onkologie Heidelberg
Locations (61):
- Germany (61):
  - Klinikum Sindelfingen-Böblingen gGmbH, Böblingen, Baden-Wurttemberg
  - Klinik für Frauenheilkunde, Universitätsklinikum Freiburg, Freiburg im Breisgau, Baden-Wurttemberg
  - NCT Heidelberg, Heidelberg, Baden-Wurttemberg
  - ViDia Christliche Kliniken Karlsruhe, Karlsruhe, Baden-Wurttemberg
  - Praxisklinik am Rosengarten, Mannheim, Baden-Wurttemberg
  - medius Klinik Nürtingen, Nürtingen, Baden-Wurttemberg
  - Universitätsfrauenklinik Tübingen, Tübingen, Baden-Wurttemberg
  - Universitätsfrauenklinik Ulm, Ulm, Baden-Wurttemberg
  - Gesundheitszentrum St. Marien GmbH, Amberg, Bavaria
  - Anregiomed gKK Klinikum Ansbach Brustzentrum Westmittelfranken, Ansbach, Bavaria
  - Hämatologische-onkologische Praxis, Augsburg, Bavaria
  - Klinikum Augsburg, Augsburg, Bavaria
  - Sozialstiftung Bamberg Klinikum am Bruderwald, Bamberg, Bavaria
  - Klinikum Bayreuth, Bayreuth, Bavaria
  - DONAUISAR Klinikum, Deggendorf, Bavaria
  - Onkologisches Zentrum Donauwörth, Donauwörth, Bavaria
  - Rottal-Inn-Kliniken GmbH, Eggenfelden, Bavaria
  - Universitätsfrauenklinik Erlangen, Erlangen, Bavaria
  - Klinikum Fürth, Fürth, Bavaria
  - MVZ am Klinikum Aschaffenburg - Zweigpraxis für Hämatologie und Onkologie, Hösbach, Bavaria
  - Onkologie Elisenhof, München, München, Bavaria
  - Klinikum der Universität München Frauenklinik, München, Bavaria
  - Frauenklinik und Poliklinik der Technischen Universität München, München, Bavaria
  - Caritas-Krankenhaus St. Josef, Regensburg, Bavaria
  - Universitätsklinikum Würzburg, Würzburg, Bavaria
  - Praxis für Frauenheilkunde und Geburtshilfe, Fürstenwalde, Brandenburg
  - Ruppiner Kliniken GmbH, Hochschulklinikum der Med. Hochschule Brandenburg, Neuruppin, Brandenburg
  - Immanuel Klinik und Poliklinik Rüdersdorf GmbH, Rüdersdorf, Brandenburg
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg, Hamburg
  - Onkologie Lerchenfeld, Hamburg, Hamburg
  - Klinikum Darmstadt Frauenklinik, Darmstadt, Hesse
  - Centrum für Hämatologie und Onkologie Bethanien, Frankfurt am Main, Hesse
  - Klinikum Kassel GmbH, Kassel, Hesse
  - Gemeinschaftspraxis für Hämatologie und Onkologie, Langen, Hesse
  - Lahn-Dill-Kliniken GmbH Klinikum Wetzlar, Wetzlar, Hesse
  - Niels-Stensen-Kliniken, Georgsmarienhütte, Lower Saxony
  - Onkologische Schwerpunktpraxis Leer-Emden, Leer, Lower Saxony
  - g.SUND Gynäkologie Kompetenzzentrum Stralsund, Stralsund, Mecklenburg-Vorpommern
  - Uniklinik RWTH Aachen, Aachen, North Rhine-Westphalia
  - Gynäkologie und Geburtshilfe im medizinischen Zentrum Bonn, Bonn, North Rhine-Westphalia
  - Marienhospital, Bottrop, North Rhine-Westphalia
  - Universitätsfrauenklinik Düsseldorf, Düsseldorf, North Rhine-Westphalia
  - Kliniken Essen-Mitte, Essen, North Rhine-Westphalia
  - Herne, North Rhine-Westphalia
  - Institut für Versorgungsforschung in der Onkologie GbR, Koblenz, North Rhine-Westphalia
  - St. Vincenz-Krankenhaus GmbH, Paderborn, North Rhine-Westphalia
  - Praxis Onkologie und Hämatologie, Recklinghausen, North Rhine-Westphalia
  - Gesellschaft für Medizinische Studien Würselen, Würselen, North Rhine-Westphalia
  - Schwerpunktpraxis für Hämatologie und Onkologie, Kaiserslautern, Rhineland-Palatinate
  - Institut für Versorgungsforschung, Mayen, Rhineland-Palatinate
  - Klinikum Chemnitz gGmbH, Chemnitz, Saxony
  - Universitätsklinik Dresden, Dresden, Saxony
  - Universitäres Krebszentrum Leipzig, Leipzig, Saxony
  - Kreiskrankenhaus Torgau, Torgau, Saxony
  - Universitätsklinikum Halle (Saale), Halle, Saxony-Anhalt
  - Klinik für Gynäkologie und Geburtshilfe, Kiel, Schleswig-Holstein
  - Universitätsklinikum Schleswig-Holstein, Lübeck, Schleswig-Holstein
  - Charité, Berlin, State of Berlin
  - MediOnko-Institut GbR, Berlin, State of Berlin
  - Klinik für Gynäkologie und Geburtshilfe, Helios Kliniken, Berlin, State of Berlin
  - medius KLINIKEN gGmbH, medius KLINIK Ostfildern-Ruit, Ostfildern

REFERENCES:
- [Derived] Muller V, Hein A, Hartkopf AD, Fasching PA, Kolberg HC, Hadji P, Tesch H, Haberle L, Ettl J, Luftner D, Wallwiener M, Beckmann MW, Schneeweiss A, Belleville E, Uhrig S, Wimberger P, Hielscher C, Meyer J, Wurmthaler LA, Kurbacher CM, Wuerstlein R, Untch M, Janni W, Taran FA, Lux MP, Wallwiener D, Brucker SY, Fehm TN, Michel LL. Occurrence and characteristics of patients with de novo advanced breast cancer according to patient and tumor characteristics - A retrospective analysis of a real world registry. Eur J Cancer. 2022 Sep;172:13-21. doi: 10.1016/j.ejca.2022.05.015. Epub 2022 Jun 18. PMID 35728342
- [Derived] Hein A, Hartkopf AD, Emons J, Lux MP, Volz B, Taran FA, Overkamp F, Hadji P, Tesch H, Haberle L, Ettl J, Luftner D, Wurmthaler LA, Wallwiener M, Muller V, Beckmann MW, Belleville E, Wimberger P, Hielscher C, Kurbacher CM, Wuerstlein R, Thomssen C, Untch M, Fasching PA, Janni W, Fehm TN, Wallwiener D, Brucker SY, Schneeweiss A, Kolberg HC. Prognostic effect of low-level HER2 expression in patients with clinically negative HER2 status. Eur J Cancer. 2021 Sep;155:1-12. doi: 10.1016/j.ejca.2021.06.033. Epub 2021 Jul 23. PMID 34311211
- [Derived] Huebner H, Kurbacher CM, Kuesters G, Hartkopf AD, Lux MP, Huober J, Volz B, Taran FA, Overkamp F, Tesch H, Haberle L, Luftner D, Wallwiener M, Muller V, Beckmann MW, Belleville E, Ruebner M, Untch M, Fasching PA, Janni W, Fehm TN, Kolberg HC, Wallwiener D, Brucker SY, Schneeweiss A, Ettl J. Heregulin (HRG) assessment for clinical trial eligibility testing in a molecular registry (PRAEGNANT) in Germany. BMC Cancer. 2020 Nov 11;20(1):1091. doi: 10.1186/s12885-020-07546-1. PMID 33176725
- See also: Biomarkers in Patients with Metastatic Breast Cancer and the PRAEGNANT Study Network — https://www.thieme-connect.de/products/ejournals/html/10.1055/s-0034-1396215